CLINICAL TRIAL: NCT05172193
Title: A Phase II Non-Randomized Open Labelled Clinical Trial to Evaluate the Safety & Immunogenicity of SARS-COV-2 Vaccine (Vero Cell) Inactivated as A Booster Dose
Brief Title: Safety & Immunogenicity of Booster SARS-CoV-2 Vaccine (Vero Cell)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PT. Kimia Farma (Persero) Tbk (Industry)
Responsible Party: Principal Investigator, Prenali Dwisthi Sattwika, Principal Investigator, Gadjah Mada University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BOOST-VC-0221
Record Dates: First submitted 2021-12-23; First posted 2021-12-29 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: COVID-19
Keywords: COVID-19; Booster; Verocell Inactivated Vaccine; Immunogenicity; Safety
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Intervention Model Description: This is a phase 2, non-randomized, open-label, clinical trial to evaluate the safety and immunogenicity of SARS-COV-2 Vaccine (Vero Cell) Inactivated up to 6 months post booster dose and a sub cohort study among vaccine arm to evaluate immunogenicity up to 12 months post booster dose in adults aged 18 years old and above who have received the 2 prime doses of one of SARSCOV-2 Vaccines (Vero Cell inactivated-Sinopharm SARS-COV-2 Vaccine, CoronaVac SARSCOV-2 Vaccine, or AstraZeneca SARS-COV-2 Vaccine) authorized for emergency use (EUA) in Indonesia.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SARS-COV-2 Vaccine (Vero Cell-Sinopharm) Inactivated (Experimental): One booster dose 0.5 mL IM injection of SARS-COV-2 Vaccine (Vero Cell) Inactivated
  Interventions: Biological: SARS-COV-2 Vaccine (Vero Cell-Sinopharm) Inactivated

INTERVENTIONS:
Biological: SARS-COV-2 Vaccine (Vero Cell-Sinopharm) Inactivated — SARS-CoV-2 vaccine (Vero cell) inactivated developed by Beijing Bio-Institute Biological Products Co., Ltd, can induce active immunity and prevent diseases caused by the SARS-CoV-2 virus by producing neutralizing antibody. The inactivated SARSCoV-2 Vaccine (Vero cell) is prepared by inoculating Verda Reno cells (Vero cell) with SARS-CoV-2 HB02 strain, culturing, harvesting, inactivating, clarifying, concentrating, purifying and adding aluminum hydroxide adjuvant.

SUMMARY:
The 2019 Coronavirus disease outbreak (COVID-19) was first reported at the end of 2019 in Wuhan China as a severe acute respiratory syndrome coronavirus 2 (SARSCoV-2) infection. In less than a year, SARS-CoV-2 infection has become a pandemic and spread to almost all countries in the world, including Indonesia. World Health Organization data states that there are 4,240,479 confirmed cases of SARS-CoV-2 in Indonesia until 25 October 2021 with a death rate of 143,235 (WHO, 2021a).

The Indonesian National Agency of Drug and Food Control (NA-DFC) has issued an Emergency Use Authorization for several SARS-COV-2 Vaccines, including the SARS-CoV-2 vaccine (Vero cell) inactivated produced by Sinopharm (BPOM, 2021). Clinical data that the actual immune responses decrease after several months are continuously being reported (Marmot et al., 2021), and the decrease of vaccine efficacy due to the appearance of variants is also known (Abu-Raddad et al., 2021; Lopez Bernal et al., 2021). These potential risks suggest the need for a booster dose or periodic booster doses of the SARS-COV-2 Vaccine. In fact, there is a study result given several months after vaccination, which leads to the generation of a higher immune responses (Pan H et al., 2021). Booster dose of SARS-COV-2 Vaccine will either induce a high level of antibody responses against original strain, or enhance the broadly formed T cell immunity regardless of mutant strain to improve individual protection.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males or females aged 18 years and above at the time of consent.
2. Participants who provide a voluntarily consent to participate in the study and sign the consent form.
3. Participants who have previously received homologous 2-dose of SARS-COV-2 Vaccine (either Vero Cell inactivated-Sinopharm SARS-COV-2 Vaccine, CoronaVac SARS-COV-2 Vaccine, or Cominarty/Pfizer mRNA COVID-19 Vaccine) authorized for emergency use, between 6 to 12 months post second prime vaccine dose prior to Day 1.
4. Participants who have negative results for swab SARS-COV-2 rapid antigen test.

Exclusion Criteria:

1. Participants who are unable to follow clinical and follow-up procedures.
2. Participants with acute fever with temperature above 38℃, coughing, breathing difficulty, chills, muscle ache, headache, sore throat, loss of smell, or loss of taste within 72 hours prior to the dosing.
3. Participants with a history of PCR-confirmed SARS-CoV-2 infection in the last 90 days prior to dosing.
4. Female who are pregnant or breastfeeding.
5. Participants with a history of hypersensitivity or allergic reactions including anaphylaxis.
6. Participants with immune dysfunction, including immunodeficiency disorder, or family history of such conditions, except HIV-positive participants in stable/well-controlled condition.
7. Participants who received chronic administration (defined as more than 14 continuous days) of immunosuppressant medication such as immunomodulator, immune-modifying drug, immunoglobulin, immunotherapy, chemotherapy, systemic corticosteroid, etc. except topical steroids or short-term oral steroids (course lasting ≤ 14 days), or blood-derived products in the last 90 days prior to dosing.
8. Participants with a current clinically significant chronic and unstable cardiovascular, endocrine, gastrointestinal, hepatic (including hepatitis B and C), renal, neurological, respiratory, psychiatric or other medical disorders not excluded by other exclusion criteria , that are assessed by the investigator as being clinically unstable within the prior 90 days as evidenced by:

   1. Hospitalization for the condition, including day surgical interventions
   2. New significant organ function deterioration
   3. Needing addition of new treatments or major dose adjustments of current treatments (mild or moderate well-controlled comorbidities are allowed)
9. Participants with hemophilia or people using anticoagulants who are at a risk of serious bleeding from IM injection.
10. Participants with a current dependent on antipsychotic drugs and narcotic analgesics, or suspected of alcohol or drug dependency.
11. Participants who have received or plans to receive other vaccination(s) within 28 days prior to or during study duration (except for influenza vaccine which is not allowed within 14 days before, or 4 weeks after final dose of IP).
12. Participants who have received or have plans to receive other investigational drug(s) while participating in another clinical study or bioequivalence study within 28 days prior to vaccination. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-12-31 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
The geometric mean titer (GMT) of anti-SARS-CoV-2 neutralizing antibody at 14 and 28 days | Within 28 days after one booster dose
  To evaluate the immunogenicity at 14 and 28 days after one booster dose of 0.5 mL intramuscular (IM) injection of SARS-COV-2 Vaccine (Vero Cell) Inactivated compared to placebo in participants who had received second dose of SARS-CoV-2 prime vaccine at least 6 months
The geometric mean fold rise (GMFR) of anti-SARS-CoV-2 neutralizing antibody at 14 and 28 days | Within 28 days after one booster dose
  To evaluate the immunogenicity at 14 and 28 days after one booster dose of 0.5 mL intramuscular (IM) injection of SARS-COV-2 Vaccine (Vero Cell) Inactivated compared to placebo in participants who had received second dose of SARS-CoV-2 prime vaccine at least 6 months
The geometric mean titer (GMT) of anti-spike protein receptor binding domain (sRBD) immunoglobulin G (IgG) antibody at 14 and 28 days | Within 28 days after one booster dose
  To evaluate the immunogenicity at 14 and 28 days after one booster dose of 0.5 mL intramuscular (IM) injection of SARS-COV-2 Vaccine (Vero Cell) Inactivated compared to placebo in participants who had received second dose of SARS-CoV-2 prime vaccine at least 6 months
The geometric mean fold rise (GMFR) of anti-spike protein receptor binding domain (sRBD) immunoglobulin G (IgG) antibody at 14 and 28 days | Within 28 days after one booster dose
  To evaluate the immunogenicity at 14 and 28 days after one booster dose of 0.5 mL intramuscular (IM) injection of SARS-COV-2 Vaccine (Vero Cell) Inactivated compared to placebo in participants who had received second dose of SARS-CoV-2 prime vaccine at least 6 months

SECONDARY OUTCOMES:
The geometric mean titer (GMT) of anti-SARS-CoV-2 neutralizing antibody at 90, 180, and 360 days | At 90, 180, and 360 days after one booster
  To evaluate the immunogenicity at 90, 180, and 360 days after one booster dose 0.5 mL IM injection of SARS-COV-2 Vaccine (Vero Cell) Inactivated compared to placebo in participants who had received second dose of SARS-CoV-2 prime vaccine at least 6 months
The geometric mean fold rise (GMFR) of anti-SARS-CoV-2 neutralizing antibody at 90, 180, and 360 days | At 90, 180, and 360 days after one booster
  To evaluate the immunogenicity at 90, 180, and 360 days after one booster dose 0.5 mL IM injection of SARS-COV-2 Vaccine (Vero Cell) Inactivated compared to placebo in participants who had received second dose of SARS-CoV-2 prime vaccine at least 6 months
The geometric mean titer (GMT) of anti-spike protein receptor binding domain (sRBD) immunoglobulin G (IgG) antibody at 90, 180, and 360 days | At 90, 180, and 360 days after one booster
  To evaluate the immunogenicity at 90, 180, and 360 days after one booster dose 0.5 mL IM injection of SARS-COV-2 Vaccine (Vero Cell) Inactivated compared to placebo in participants who had received second dose of SARS-CoV-2 prime vaccine at least 6 months
The geometric mean fold rise (GMFR) of anti-spike protein receptor binding domain (sRBD) immunoglobulin G (IgG) antibody at 90, 180, and 360 days | At 90, 180, and 360 days after one booster
  To evaluate the immunogenicity at 90, 180, and 360 days after one booster dose 0.5 mL IM injection of SARS-COV-2 Vaccine (Vero Cell) Inactivated compared to placebo in participants who had received second dose of SARS-CoV-2 prime vaccine at least 6 months
To proportion of solicited adverse events within 7 days after one booster dose | Within 7 days after one booster
  To evaluate the safety profile of one booster dose 0.5 mL IM injection of SARSCOV-2 Vaccine (Vero Cell) Inactivated in participants who had received second dose of SARS-CoV-2 prime vaccine at least 6 months
To proportion of unsolicited adverse events within 28 days after one booster dose | Within 28 days after one booster
  To evaluate the safety profile of one booster dose 0.5 mL IM injection of SARSCOV-2 Vaccine (Vero Cell) Inactivated in participants who had received second dose of SARS-CoV-2 prime vaccine at least 6 months
To proportion of clinically significant abnormal liver function (AST, ALT, Total Bilirubin) at 14 days and 28 days | Within 28 days after one booster
  To evaluate the safety profile of one booster dose 0.5 mL IM injection of SARSCOV-2 Vaccine (Vero Cell) Inactivated in participants who had received second dose of SARS-CoV-2 prime vaccine at least 6 months
To proportion of serious adverse events within 180 days after one booster dose | Within 180 days after one booster
  To evaluate the safety profile of one booster dose 0.5 mL IM injection of SARSCOV-2 Vaccine (Vero Cell) Inactivated in participants who had received second dose of SARS-CoV-2 prime vaccine at least 6 months

OTHER OUTCOMES:
To proportion of symptomatic PCR-confirmed SARS-CoV-2 infection within 90 and 180 days after one booster dose | Within 180 days after one booster
  To evaluate proportion of symptomatic PCR-confirmed SARS-CoV-2 infection after one booster dose 0.5 mL IM injection of SARS-COV-2 Vaccine (Vero Cell) Inactivated compared to placebo in participants who had received second dose of SARS-CoV-2 prime vaccine at least 6 months

CONTACTS AND LOCATIONS:
Locations (7):
- Indonesia (7):
  - Universitas Udayana Hospital, Badung, Bali
  - Bali Mandara Hospital, Denpasar, Bali
  - Kimia Farma Soetomo Clinic and Laboratorium, Semarang, Central Java
  - JIH Hospital, Sleman, D.I. Yogyakarta
  - Kimia Farma Adisucipto Clinic and Laboratorium, Yogyakarta, D.I. Yogyakarta
  - Kimia Farma Diponegoro Clinic and Laboratorium, Bandung, West Java
  - Kimia Farma Radio Dalam Clinic and Laboratorium, Jakarta

IPD SHARING:
Plan to Share IPD: No